CLINICAL TRIAL: NCT01748708
Title: Evaluating the Efficacy of Magnetic Seizure Therapy in Treatment Resistant Depression.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol has undergone significant changes and the investigator feels that it is reasonable to submit a new protocol for review and approval.
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080-2012
Record Dates: First submitted 2012-12-11; First posted 2012-12-12 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Depressive Disorder
Keywords: Magnetic seizure therapy; Electroconvulsive therapy; Treatment resistant depression; Treatment resistance; Randomized controlled trial
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic seizure therapy (Experimental)
  Interventions: Device: Magnetic seizure therapy
- Electroconvulsive therapy (Active Comparator)
  Interventions: Device: Electroconvulsive therapy

INTERVENTIONS:
Device: Magnetic seizure therapy — 100% machine output at 100 Hz, with coil directed over frontal brain regions, until adequate seizure achieved. Treatments will be administered 3 times per week, up to a maximum of 15 treatments. If subjects fail to achieve the pre-defined criteria of remission at that point, they will be considered non-remitters and will exit the study.
  Other Names: MagPro MST (Tonica Elektronik A/S, Denmark)
  Arms: Magnetic seizure therapy
Device: Electroconvulsive therapy — ECT treatments will be administered 3 times per week using the MECTA spECTrum 5000Q. Subjects will be treated with an ultrabrief (0.3ms) pulse with a bilateral placement at 6 times the seizure threshold, up to a maximum of 15 treatments. If subjects fail to achieve the pre-defined criteria of remission at that point, they will be considered non-remitters and will exit the study.
  Other Names: MECTA spECTrum 5000Q
  Arms: Electroconvulsive therapy

SUMMARY:
Electroconvulsive therapy (ECT) has unparalleled efficacy in treating severe depression that is resistant to common modalities of treatment, such as antidepressant medication. Although treatment with ECT has benefited many individuals with treatment resistant depression (rates as high as 50-75%), its more widespread use is hindered by the social stigma associated with the treatment, as well as by its significant cognitive side effects. Moreover, ECT cannot be precisely targeted, since it produces a widespread activation of the brain surface, in turn, affecting many different functional areas. Magnetic seizure therapy (MST) is currently being investigated as an alternative to ECT, as it is more focused to one area of the brain. Rather than applying electrical stimuli to induce a seizure, as is done in ECT, MST uses repetitive magnetic stimulation to produce the seizure. Preliminary research suggests that MST can result in therapeutic effects comparable to those produced by ECT, but without the negative side effects on cognition. The proposed study is a randomized, controlled trial, in which the efficacy and side effect profile of MST will be compared to those of ECT. If successful, the results of this study may lead to increased treatment availability and accessibility, as well as lessen the substantial health care costs associated with treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* inpatients or outpatients
* voluntary and competent to consent to treatment
* DSM-IV diagnosis of major depressive disorder, single or recurrent, without psychotic features
* have failed to achieve a clinical response to adequate treatment trials of at least two antidepressants (with adequacy established according to a predefined criterion on the Antidepressant Treatment History Form (ATHF)) or have been unable to tolerate at least two antidepressants
* have a baseline HRSD-24 score ≥ 21
* are considered to be appropriate to receive ECT as assessed by an ECT attending psychiatrist and an anaesthesiologist
* are agreeable to keeping their current antidepressant treatment constant through the duration of the study
* are able to adhere to the intervention schedule
* meet the MST safety criteria
* are on a medically acceptable form of birth control if a woman of child-bearing potential
* are a resident of Canada

Exclusion Criteria:

* have a history of DSM-IV substance dependence or abuse within the past three months
* have a concomitant major unstable medical illness
* are acutely suicidal with imminent intent
* are pregnant or intend to get pregnant during the study
* have a DSM-IV confirmed diagnosis of bipolar disorder, any psychotic disorder, obsessive compulsive disorder, or post-traumatic stress disorder (current or within the last year)
* have a DSM-IV diagnosis of borderline personality disorder as assessed by a study investigator
* have possible or probable dementia
* have failed a course of ECT within the current depressive episode
* have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or cognitive impairment (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis, head trauma with loss of consciousness for greater than or equal to five minutes)
* present with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease)
* have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* require a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT
* have an inability to communicate in English fluently enough to complete the neuropsychological tests
* have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression, 24-item (HRSD-24) | Change from baseline in HRSD-24 score at date of symptom remission or date of the 15th treatment, whichever comes first, assessed up to 6 months.
  The HRSD-24 is a semi-structured, clinician-administered scale used to assessed the severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Z. Jeffrey Daskalakis, MD, PhD., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research/Pages/research.aspx